CLINICAL TRIAL: NCT00689520
Title: Phase IV, Randomized, Open-Label Trial Comparing Long-Term Subcutaneous Low-Molecular Weight Heparin With Oral Anticoagulant Therapy in the Treatment of Deep Venous Thrombosis
Brief Title: Long-Term Low-Molecular-Weight Heparin Versus Oral Anticoagulants in Deep Venous Thrombosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: LEO Pharma (Industry)
Responsible Party: Romera, Antonio MD, Department of Vascular Surgery. Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV1/01; CV1/01
Record Dates: First submitted 2008-05-28; First posted 2008-06-03 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-05

CONDITIONS: Venous Thromboembolism
Keywords: Venous thromboembolism; low molecular weight heparin; Vitamin K antagonist; Longterm
MeSH Terms: conditions — Venous Thromboembolism | interventions — Tinzaparin; Acenocoumarol; acarboxyprothrombin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tinzaparin (Experimental): tinzaparin (Innohep®) subcutaneously in a fixed dose of 175 IU anti-Xa/kg of body weight once daily for 6 months.
  Interventions: Drug: tinzaparin
- acenocoumarol (Active Comparator): tinzaparin for 1 weeks followed by acenocoumarol for 6 months
  Interventions: Drug: acenocoumarol

INTERVENTIONS:
Drug: tinzaparin — tinzaparin (Innohep®) subcutaneously in a fixed dose of 175 IU anti-Xa/kg of body weight once daily for 6 months
  Other Names: innohep
  Arms: tinzaparin
Drug: acenocoumarol — tinzaparin subcutaneously 175 IU anti-Xa/kg of body weight once daily for 7 days followed by acenocoumarol for 6 months
  Other Names: Vitamin K antagonists
  Arms: acenocoumarol

SUMMARY:
The purpose of this study is to evaluate whether low-molecular-weight heparin could be equally or more effective than oral anticoagulation in the long-term treatment of deep venous thrombosis.

DETAILED DESCRIPTION:
The open-label prospective randomized clinical trial compares subcutaneous LMWH (tinzaparin)administered for 6 months versus initial treatment using subcutaneous LMWH followed by oral anticoagulants given for a similar period of time in patients with proximal venous thrombosis.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive, symptomatic patients with a first or recurrent episode of acute proximal-vein thrombosis of the lower limbs.
* either sex and over 18 years of age
* referred to the Vascular Surgery Department of the hospital
* onset of symptoms less than 2 weeks
* documented by compression ultrasonography,

Exclusion Criteria:

* received heparin, low-molecular-weight heparin or oral anticoagulant therapy for more than 2 days for the present disease
* pulmonary embolism requiring thrombolytic therapy
* Need of surgical thrombectomy or vena cava interruption
* receiving oral anticoagulant treatment or antiplatelet agents for other conditions
* contraindication to anticoagulant treatment (active bleeding, severe blood pressure or allergy to the study drugs)
* platelet count lower than 100x103 /μl or hemoglobin concentration lower than 7 g/dl or history of heparin-associated thrombocytopenia
* severe renal failure necessitating dialysis
* pregnancy
* lumbar puncture within the previous 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2002-01; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic recurrent venous thromboembolism | 12 months

SECONDARY OUTCOMES:
Occurrence of major bleeding | 6 month treatment interval

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Romera, MD, Study Chair — Hospital Universitari de Bellvitge; Antoni Romera, MD, Principal Investigator — Hospital Universitari de Bellvitge; Oriol Lapiedra, MD, Principal Investigator — Hospital Creu Roja de l'Hospitalet
Locations (2):
- Spain (2):
  - Vascular surgery service. Hospital Creu Roja de l'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Department of Vascular Surgery. Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona